CLINICAL TRIAL: NCT04683640
Title: Sleep, Pain and Aging: Potential Underlying Mechanisms
Brief Title: Latent Aging Mechanisms in Pain and Sleep
Acronym: LAMPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Thorne HealthTech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB202000105-N; P30AG059297 (NIH)
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — gamma-Aminobutyric Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daily Oral GABA (Experimental): You will take, by mouth, 2 pills of GABA (500 mg) (Capsule 250mg) daily at home for 4 weeks
  Interventions: Dietary Supplement: GABA
- Daily Placebo (Placebo Comparator): You will take, by mouth, 2 pills of Placebo daily at home for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: GABA — Daily oral GABA for 4 weeks
  Other Names: Gamma aminobutyric acid
  Arms: Daily Oral GABA
Drug: Placebo — Daily oral Placebo for 4 weeks
  Arms: Daily Placebo

SUMMARY:
Chronic pain is a serious public health problem in older adults depending on the pain condition, and the capacity to sleep properly changes with age. Given the potential mechanistic role of GABA (gamma-aminobutyric acid) in both conditions, based on our preliminary data, this proposal will determine the effect of oral GABA administration in sleep quality and pain in older adults with chronic pain and sleep disorders as well as to characterize the potential neurobiological mechanisms involved in both illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Older adults 45 years of age or older who experienced pain of at least moderate intensity (>5/10 pain intensity ratings) on more days than not during the past three months, and who also reported poor sleep quality (>5 PSQI scores) will be considered for participation.

Exclusion Criteria:

1. serious psychiatric conditions (e.g., schizophrenia, major depression, bipolar disorder;
2. history of alcohol/drug abuse;
3. Alzheimer, Parkinson, Epilepsy and other known intra-cerebral pathology and neurological conditions;
4. significant cognitive impairment as evidenced by the Modified Mini-Mental State Examination [3MS] score ≤ 77;
5. hospitalizations for mental health reasons in the past year;
6. chronic/current use of narcotic medications;
7. serious systemic (uncontrolled diabetes self-reported HA1C>7), (uncontrolled hypertension > 155/90 mm Hg) and rheumatic disorders (i.e., rheumatoid arthritis, systemic lupus erythematosus, fibromyalgia, HIV);
8. arterial hypotension;
9. digestive tract diseases;
10. major medical surgery in the past two months, history of brain surgery or any serious brain condition like aneurysm, stroke, or seizures;
11. excessive anxiety regarding protocol procedures;
12. Inability to consent for study participation;
13. Ingestion of sleep medications including those with zolpidem (Ambien and others) and eszopiclone (Lunesta and others);
14. Neuropathic pain medications including anticonvulsants and antidepressants;
15. Allergies or sensitivity to GABA or its ingredients cellulose' gelatin (capsule)' magnesium silicate' vegetable stearate and silica or to the placebo or its ingredients: calcium laurate, hypromellose capsule, magnesium (citrate), microcrystalline cellulose;
16. currently taking barbiturate and benzodiazepine and baclofen;
17. MRI contraindications including large pieces of metal in the body/face/neck and claustrophobia;
18. current cancer diagnosis unless determined no evidence of disease or in remission for at least two years, and
19. pregnancy

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yenisel Cruz-Almeida, MSPH, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants completed a screening visit and provided written informed consent before randomization. No run-in or washout phases were implemented before treatment initiation.
Groups:
- PLACEBO: Participants self-administered Placebo (microcrystalline cellulose) capsules (two capsules) daily at home at 08:00 pm for 4 weeks.
- GABA: Participants self-administered PharmaGABA-250 (gamma-aminobutyric acid 250 mg/cap) 500 mg orally (two 250 mg capsules) daily at home at 08:00 pm for 4 weeks.
Period: Overall Study
Arm/Group | PLACEBO | GABA
Started | 15 | 18
Completed | 13 | 17
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for participants who completed the baseline assessment and had complete data for the variables analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO | GABA | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 12 | 12 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 15 | 18 | 33
The Pittsburgh Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: Units on a scale (0-21).] — The Pittsburgh Sleep Quality Index (PSQI) is a validated self-reported questionnaire designed to assess sleep quality and disturbances over the past month. The PSQI total score ranges from 0 to 21, with higher scores indicating worse sleep quality. A total score greater than 5 indicates poor sleep quality.
  Units on a scale (0-21). | 11.20 (4.18) | 9.78 (3.02) | 10.43 (3.59)

OUTCOME MEASURES:

1. Primary Outcome: The Pittsburgh Sleep Quality Index (PSQI): PSQI Total Score at Baseline
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over the past month. It consists of 19 items grouped into seven components. Each component is scored from 0 to 3, and the component scores are summed to yield a global total score ranging from 0 to 21. Higher scores indicate worse sleep quality. A total score greater than 5 is typically used to distinguish poor sleepers from good sleepers.
Time Frame: PSQI was administered at baseline
Population: Baseline characteristics for the Pittsburgh Sleep Quality Index (PSQI) are reported for participants who completed the baseline assessment and had complete PSQI data.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 15 | 18
Score on scale | 11.20 (4.18) | 9.78 (3.02)

2. Primary Outcome: The Pittsburgh Sleep Quality Index (PSQI): PSQI Total Score at Post-Intervention
Description: as for outcome 1
Time Frame: PSQI was administered immediately after completing the 4-week intervention
Population: The number of participants analyzed post-intervention differs from the baseline assessment due to missing data. Two participants in Group A did not complete the PSQI at the post-intervention time point and were therefore excluded from the post-intervention analysis. All other participants included had complete data.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 13 | 18
Score on scale | 8.08 (3.59) | 7.89 (3.23)

3. Primary Outcome: Verbal Descriptor Scale (VDS) at Baseline
Description: The Verbal Descriptor Scale (VDS) is a validated self-report measure of pain intensity, commonly used in older adults. Participants are asked to select the descriptor that best represents their current pain level from six options: No pain, Mild, Moderate, Severe, Very severe, and Worst possible pain. Each descriptor corresponds to a numeric value from 0 to 5, with higher scores indicating greater pain intensity.
Time Frame: VDS was administered at baseline
Population: The analysis population for the Verbal Descriptor Scale (VDS) at baseline includes all participants who were assigned to Group A (n=15) and Group B (n=18), as all completed the baseline assessment.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 15 | 18
Scores on a scale | 2.00 [1 to 2] | 1.50 [1 to 2]

4. Primary Outcome: Verbal Descriptor Scale (VDS) at Post-Intervention
Description: as for outcome 3
Time Frame: VDS was administered immediately after completing the 4-week intervention
Population: The number of participants analyzed post-intervention differs from the baseline assessment due to missing data. Two participants in Group A did not complete the VDS at the post-intervention time point and were therefore excluded from the post-intervention analysis. All other participants included had complete data.
Measure: Median (Inter-Quartile Range); unit: Score on scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 13 | 18
Score on scale | 1 [0.50 to 2] | 1 [1 to 2]

5. Primary Outcome: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) at Baseline
Description: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a validated self-report questionnaire that assesses pain, stiffness, and physical function in individuals with musculoskeletal conditions. It includes 24 items scored on a 5-point Likert scale (0 = none to 4 = extreme), producing subscale scores and a total score. The total WOMAC score ranges from 0 to 96, with higher scores indicating worse symptoms and functional limitations.
Time Frame: WOMAC was administered at baseline.
Population: The analysis population for the WOMAC at baseline includes all participants who were assigned to Group A (n=15) and Group B (n=18), as all completed the baseline assessment.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 15 | 18
Score on scale | 33.83 (18.98) | 34.77 (18.61)

6. Primary Outcome: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) at Post-Intervention
Description: as for outcome 5
Time Frame: WOMAC was administered after completing the 4-week intervention
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 15 | 18
Score on scale | 22.92 (17.98) | 34.87 (19.41)

7. Secondary Outcome: Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) Total Score at Baseline
Description: The Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) is a validated 22-item self-report instrument that assesses the multidimensional experience of pain. Items are grouped into four subscales-continuous, intermittent, neuropathic, and affective pain-and each item is rated from 0 (no pain) to 10 (worst possible pain) based on pain intensity over the past week. The total score is calculated as the average of all 22 item scores, with higher scores indicating greater pain severity.
Time Frame: Baseline
Population: The number of participants analyzed differs from the number of participants assigned to the group due to missing data. One participant in Group B did not complete the SF-MPQ-2 at baseline time point and was, therefore, excluded from the baseline analysis. All other participants included had complete data.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 15 | 17
Score on scale | 2.41 (1.63) | 2.21 (1.62)

8. Secondary Outcome: Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) Total Score at Post-Intervention
Description: as for outcome 7
Time Frame: Immediately post-intervention (4 weeks)
Population: The number of participants analyzed post-intervention differs from the baseline assessment due to missing data. Two participants in Group A did not complete the SF-MPQ-2 at the post-intervention time point and were, therefore, excluded from the post-intervention analysis. All other participants included had complete data.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 13 | 18
Score on scale | 1.43 (1.14) | 1.77 (1.36)

9. Secondary Outcome: Pain Detect at Baseline
Description: The PainDETECT Questionnaire is a validated self-report instrument used to assess the likelihood of a neuropathic pain component in individuals with chronic pain. It includes 9 items that assess pain intensity, pain patterns, and sensory descriptors. The total score ranges from -1 to 38, with higher scores indicating a greater probability of neuropathic pain. A score ≥19 suggests likely neuropathic pain, 13-18 indicates possible neuropathic pain, and ≤12 suggests that neuropathic pain is unlikely.
Time Frame: Baseline
Measure: Median (Standard Deviation); unit: Score on scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 15 | 18
Score on scale | 9.23 (5.70) | 9.39 (6.89)

10. Secondary Outcome: Pain Detect at Post-Intervention
Description: as for outcome 9
Time Frame: Immediately post-intervention (4 weeks)
Population: The number of participants analyzed post-intervention differs from the baseline assessment due to missing data. Two participants in Group A did not complete the Pain Detect at the post-intervention time point and were, therefore, excluded from the post-intervention analysis. All other participants included had complete data.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 13 | 18
Score on scale | 6.54 (5.17) | 8.33 (6.27)

11. Secondary Outcome: Functional Outcomes of Sleep Questionnaire - 10 Items (FOSQ-10) at Baseline
Description: The Functional Outcomes of Sleep Questionnaire-10 (FOSQ-10) is a 10-item self-report instrument that assesses the impact of excessive daytime sleepiness on daily functioning across five domains. Each item is rated on a 4-point Likert scale from 1 (extreme difficulty) to 4 (no difficulty). The total score is calculated by averaging items within each domain and summing the domain means. Total scores range from 5 to 20, with higher scores indicating better functional status and less impairment.
Time Frame: Baseline
Population: The number of participants analyzed differs from the number of participants assigned to the group due to missing data. Three participants in Group A, and two in Group B, did not complete the FOSQ-10 at the baseline time point and were, therefore, excluded from the baseline analysis. All other participants included had complete data.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 12 | 16
Score on scale | 17.54 (1.28) | 16.58 (2.84)

12. Secondary Outcome: Functional Outcomes of Sleep Questionnaire - 10 Items (FOSQ-10) at Post-Intervention
Description: as for outcome 11
Time Frame: Immediately post-intervention (4 weeks)
Population: The number of participants analyzed post-intervention differs from the baseline assessment due to missing data. Two participants in Group A did not complete the FOSQ-10 at the post-intervention time point and were therefore excluded from the post-intervention analysis. All other participants included had complete data.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 12 | 18
Score on scale | 12.60 (2.70) | 12.48 (2.65)

13. Secondary Outcome: Epworth Sleepiness Scale (ESS) at Baseline
Description: The Epworth Sleepiness Scale (ESS) is an 8-item self-report questionnaire that assesses the likelihood of dozing off or falling asleep during common daily activities. Each item is scored from 0 (would never doze) to 3 (high chance of dozing). The total score is calculated by summing the scores across all 8 items, yielding a total range of 0 to 24, with higher scores indicating greater levels of daytime sleepiness.
Time Frame: Baseline
Population: The number of participants analyzed differs from the number of participants assigned to the group due to missing data. Three participants in Group A, and two in Group B, did not complete the ESS at the baseline time point and were, therefore, excluded from the baseline analysis. All other participants included had complete data.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 12 | 16
Score on scale | 6.67 (3.03) | 8.56 (4.13)

14. Secondary Outcome: Epworth Sleepiness Scale (ESS) at Post-Intervention
Description: as for outcome 13
Time Frame: Immediately post-intervention (4 weeks)
Population: The number of participants analyzed differs from the number of participants assigned to the group due to missing data. Three participants in Group A did not complete the ESS at the post-intervention time point and were, therefore, excluded from the post-intervention analysis. All other participants included had complete data.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | PLACEBO | GABA
Number analyzed (Participants) | 12 | 18
Score on scale | 7.08 (4.44) | 7.56 (5)

ADVERSE EVENTS:
Time Frame: From the start of the intervention through 3 months post-intervention. Adverse events were actively monitored weekly during the 4-week treatment phase and followed up for an additional 3 months after study completion
Description: Adverse events in this study were defined as any unfavorable or unintended signs, symptoms, or conditions reported by participants during the study period, regardless of relatedness to the intervention.
  Adverse events were systematically assessed through weekly check-in calls during the 4-week intervention phase and continued via follow-up for 3 months post-intervention. All events reported were non-serious, local, and categorized as possibly related to the study procedures.
Arm/Group | PLACEBO | GABA
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/18
Other Adverse Events (participants affected / at risk) | 12/15 | 17/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=15) | GABA (N=18)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal/stomach pain (Gastrointestinal disorders) | 3 (3) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Balance problems (Nervous system disorders) | 0 (0) | 9 (9)
Blurred vision (Eye disorders) | 2 (2) | 5 (5)
Causing difficulty sleeping longer (Social circumstances) | 1 (1) | 0 (0)
Change in appetite (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Feelings of stress or anxiety (Psychiatric disorders) | 8 (8) | 8 (8)
Glucose high/ thirsty (Endocrine disorders) | 1 (1) | 1 (1)
Heart rate changes/palpitations (Cardiac disorders) | 2 (2) | 5 (5)
Left shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Light-headedness/vertigo (Nervous system disorders) | 6 (6) | 8 (8)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Right leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin rash/itching (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Changes in blood pressure (Vascular disorders) | 2 (2) | 1 (1)
Changes in mood (Psychiatric disorders) | 4 (4) | 6 (6)
Constipation (Gastrointestinal disorders) | 7 (7) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Drowsiness/sleepiness (Nervous system disorders) | 11 (11) | 11 (11)
Tired (General disorders) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (9)
Fatigue (General disorders) | 8 (8) | 12 (12)

LIMITATIONS AND CAVEATS:
This study was a single-site, proof-of-concept trial with a relatively small sample size, which may limit generalizability. The study remained blinded at the time of reporting; group assignments were not unmasked for outcome comparisons. Some outcome measures had missing post-intervention data, particularly in Group A, potentially impacting statistical power. The adverse event reporting table may reflect minor inconsistencies in total counts due to repeat occurrences per participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT04683640/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT04683640/ICF_001.pdf